CLINICAL TRIAL: NCT06298968
Title: Combined Therapy Using Gemcitabine and Cisplatin Chemotherapy, Lenvatinib and Adebrelimab for Patients With Advanced and Unresectable Intrahepatic Cholangiocarcinoma: a Prospective, Single-arm, Phase II Trial.
Brief Title: Combined Therapy Using Gemcitabine and Cisplatin Chemotherapy, Lenvatinib and Adebrelimab for Patients With Advanced and Unresectable Intrahepatic Cholangiocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2024-074
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: Lenvatinib; Adebrelimab; gemcitabine; cisplatin
MeSH Terms: conditions — Cholangiocarcinoma | interventions — lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined therapy using GC, Lenvatinib and Adebrelimab (Experimental): GC chemotherapy every 3 weeks,with a total of 6 cycles. Lenvatinib 8 mg once daily (QD) oral dosing. Adebrelimab 1200mg intravenously every 3 weeks.
  Interventions: Drug: combined therapy using gemcitabine and cisplatin chemotherapy, Lenvatinib and Adebrelimab

INTERVENTIONS:
Drug: combined therapy using gemcitabine and cisplatin chemotherapy, Lenvatinib and Adebrelimab — Gemcitabine (1000mg/m²) and cisplatin (25mg/m²) on day1 and 8 every 3 weeks, with a total of 6 cycles.
  Lenvatinib 8 mg once daily (QD) oral dosing, continuous use for 2 years. Adebrelimab 1200mg intravenously every 3 weeks, continuous use for 2 years.

SUMMARY:
In this phase 2 study, the investigators aim to evaluate the efficacy and safety of combined therapy using gemcitabine and cisplatin chemotherapy, Lenvatinib and Adebrelimab for patients with advanced and unresectable intrahepatic cholangiocarcinoma

DETAILED DESCRIPTION:
Most intrahepatic cholangiocarcinoma (ICC) patients are often accompanied by local or distant metastases and lose the opportunity for surgical resection. For patients with unresectable ICC who have been in stages IIIb and IV (AJCC/UICC, V2, 2018), the survival time is less than 4 months, and there is currently no standard treatment. TheGC chemotherapy (gemcitabine and cisplatin) has been used in the treatment of advanced intrahepatic cholangiocarcinoma, but the efficacy is still unsatisfactory. Lenvatinib is a small molecule multi-kinase inhibitor, the main targets including VEGFR1-3, fibroblast growth factor receptor 1-4, PDGFRα, RET(ret proto-oncogene ), KIT(KIT proto-oncogene, receptor tyrosine kinase), have anti-angiogenic effects, have been proven effective in hepatocellular carcinoma. In recent years, immunological checkpoint inhibitors (ICIs) have shown remarkable therapeutic effects in the treatment of various solid tumors. Combined with other therapies such as chemotherapy and targeted drugs is an important direction to improve the therapeutic effect of immunological checkpoint inhibitors. In this study, the investigators aim to evaluate the efficacy and safety of GC chemotherapy combined with Lenvatinib and immune checkpoint inhibitor PD-L1 antibody Adebrelimab for patients with advanced and unresectable intrahepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be required to sign an informed consent form;
2. Age 18-75 years old, male or female;
3. Eastern Cooperative Oncology Group (ECOG) fitness status score (PS score) 0-1;
4. Child-Pugh score A;
5. Histopathologically confirmed intrahepatic cholangiocarcinoma; consent to provide previously stored tumor tissue specimens or fresh biopsy tumor lesions;
6. Advanced and unresectable ICC patients;
7. The expected survival is longer than 12 weeks;
8. At least 1 measurable liver lesion or non-liver lesion (according to RECIST 1.1);
9. Functional indicators of vital organs meet the following requirements a Neutrophils ≥1.5*109/L; platelets≥100*109/L; hemoglobin≥9g/dl; serum albumin≥3g/dl; b Thyroid stimulating hormone (TSH) ≤ 1 times the upper limit of normal value(ULN), T3, T4 are in the normal range; c bilirubin ≤ 2 times ULN; Alanine aminotransferase （ALT） and Aspartate aminotransferase （AST） ≤ 2 times ULN; serum creatinine ≤ 1.5 ULN, creatinine clearance rate ≥ 60ml / min;
10. Non-lactating or pregnant women, contraception during or after 3 months of treatment.

Exclusion Criteria:

1. Pathological diagnosis of hepatocellular carcinoma, mixed liver cancer and other non-cholangiocarcinoma malignant tumor components;
2. Patients who have received previous treatment with PD1 antibody, programmed death ligand -1 （PD-L1） antibody or cytotoxic T lymphocyte-associated antigen-4 （CTLA4） antibody;
3. With other malignant tumors, except for fully treated non-melanoma skin cancer, cervical carcinoma in situ, and papillary thyroid carcinoma;
4. Active tuberculosis infection. Patients with active tuberculosis infection within 1 year prior to enrollment; had a history of active tuberculosis infection more than 1 year before enrollment, did not receive formal anti-tuberculosis treatment or tuberculosis is still active;
5. Have an active, known or suspected autoimmune disease. Subjects who require only hormone replacement therapy for hypothyroidism and skin diseases that do not require systemic therapy may be enrolled;
6. Previous interstitial lung disease, or (non-infectious) pneumonia and need oral or intravenous steroid therapy;
7. Long-term systemic hormones (dose equivalent to >10 mg prednisone/day) or any other form of immunosuppressive therapy are required. Subjects using inhaled or topical corticosteroids may be enrolled;
8. Severe cardiopulmonary and renal dysfunction;
9. Suffering from high blood pressure, and can not be well controlled by antihypertensive drugs (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg);
10. Abnormal blood coagulation (PT>14s), with bleeding tendency or receiving thrombolytic or anticoagulant therapy;
11. Hepatitis B virus （HBV） DNA>2000 copies/ml, hepatitis C virus （HCV） RNA>1000;
12. Significant clinically significant bleeding symptoms or a clear tendency to appear within 6 months prior to enrollment;
13. Active infections requiring systemic treatment;
14. Human immunodeficiency virus (HIV) positive;
15. History of psychotropic substance abuse, alcohol abuse or drug abuse;
16. Has a history of allergy to platinum;
17. Other factors that may influence the safety of the subject or the compliance of the test by the investigator. Serious illnesses (including mental illness), severe laboratory tests, or other family or social factors that require combined treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2025-02-25 (Estimated); Study Completion 2027-02-25 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From date of first dose of study drug until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to approximately 3 years
  ORR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) at the time of data cutoff as assessed by RECIST 1.1

SECONDARY OUTCOMES:
The disease control rate (DCR) | From date of first dose of study drug until disease progression, stable disease, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to approximately 3 years)
  DCR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) or stable disease (SD) at the time of data cutoff as assessed by RECIST 1.1
Duration of response (DOR) | From the first documentation of CR or PR to the first date of documentation of disease progression or death whichever occurs first (up to approximately 3 years)
  DOR is defined as the time from the first documentation of CR or PR to the date of first documentation of disease progression or death (whichever occurs first) as assessed by RECIST 1.1
The median progression free survival time (mPFS) | From date of first dose of study drug to the date of first documentation of disease progression (up to approximately 3 years)
  The progression free survival time (mPFS) defined as the time from the first study dose date to the date of first documentation of disease progression as assessed by RECIST 1.1
The median overall survival time (mOS) | From the start date of the Treatment Phase until date of death from any cause (up to approximately 3 years)
  OS is measured from the start date of the Treatment Phase (date of first study dose) until date of death from any cause. Participants who are lost to follow-up and the participants who are alive at the date of data cutoff will be censored at the date the participant was last known alive or the cut-off date, whichever comes earlier.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | From the start date of the Treatment Phase until date of death from any cause (up to approximately 3 years)
  Safety will be evaluated according to the NCI CTCAE Version 5.0. All observations pertinent to the safety of the study medication will be recorded on the CRF and included in the final report.

CONTACTS AND LOCATIONS:
Overall Officials: Jinzhang Chen, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No